CLINICAL TRIAL: NCT04688866
Title: Investigation Into the Fungal Microbiome (Mycobiome) in the Cervices of Cervical Insufficiency Patients Receiving Cerclage Treatment and Resulting in Term or Preterm Birth
Brief Title: Investigation Into the Microorganisms in Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hallym University (Other); Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Stephen Chim, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2012.243
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Cervical Insufficiency; Preterm Birth
Keywords: preterm birth; cervical insufficiency; cerclage; pessary
MeSH Terms: conditions — Uterine Cervical Incompetence; Premature Birth | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Cervical swab samples obtained comprise ample amount of DNA for PCR amplification or sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with cervical insufficiency (Cases): Pregnant women with a shortened (<25 mm) or dilated cervix in the second trimester (or late first trimester)
  Interventions: Other: Sequencing
- Pregnant women without cervical insufficiency (Controls): Pregnant women with a normal-length (>= 25 mm) and closed cervix in the second trimester (or late first trimester)
  Interventions: Other: Sequencing

INTERVENTIONS:
Other: Sequencing — This is an observational study, since the assignment of the medical intervention (e.g. cerclage or pessary) is not at the discretion of the investigator. However, cervical samples collected from both groups are subjected to amplicon sequencing for taxonomic classification of microorganisms.

SUMMARY:
Pregnant women with short cervical length (<25 mm) in second-trimester ultrasonographic assessment are at high risk for preterm birth, a major cause of perinatal mortality and morbidity worldwide. Some of these short-cervix women proceed to a more advanced stage manifested as a painless prematurely dilated cervix in the second trimester. It is not fully understood why some women have short cervical length or prematurely dilated cervix (cervical insufficiency), although evidence is mounting that there is an association between short cervical length and infection by microorganisms. The investigators hypothesize that the cervical microorganisms in pregnant women with a shortened or dilated cervix are different, compared with those in women with normal cervical length and a closed cervix.

DETAILED DESCRIPTION:
Previously, culture-dependent methods were used to detect bacterial or fungal infection, but the sensitivity was low, since not all species grew well in culture. Recently, molecular methods based on PCR amplification of the bacterial 16S ribosomal RNA (rRNA) gene or the fungal internal transcribed spacer (ITS) followed by capillary sequencing has been used to identify bacteria and fungi. However, the resolution of such capillary sequencing-based method (<100 sequencing reads/sample) is too low to capture the major collection of microorganisms in a sample. Less abundant but possibly pathogenic microorganisms associated with short cervical length remain undetectable. To address the current gap in this field, we propose to more comprehensively survey microbial communities in the cervix of pregnant women by PCR amplification of the 16S rRNA region, ITS or other genomic regions with taxonomic classification potential. This will be followed by next-generation sequencing (>40,000 sequencing reads/sample), which has been proven to capture the majority of microorganisms in a sample.

ELIGIBILITY:
Inclusion Criteria:

* Women with or without cervical insufficiency (cervical length <25 mm or dilated cervix in the second trimester or the late first trimester)

Exclusion Criteria:

* multiple pregnancies and pregnancies associated with fetal chromosomal abnormality

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women who attend preterm clinics or receive antenatal care at the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-06-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Abundances of microorganisms in the cervix | 1 year
  Abundances of microorganisms including bacteria and fungi in the cervix are measured by normalized sequencing read counts

SECONDARY OUTCOMES:
Gestational age at delivery | 1 year
Mode of delivery | 1 year
Number of participants who received cerclage or ring pessary in the current pregnancy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S Chim, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Research Laboratory, Dept of Obstetrics & Gynaecology, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No